CLINICAL TRIAL: NCT05352620
Title: Smart Box Accompanied With OT Equator Attachment in Retaining Immediately Loaded Inclined Implant Assisted Overdenture for Atrophic Maxilla
Brief Title: Smart Box With OT Equator Attachment in Retaining Implant-assisted Overdenture for the Atrophic Maxilla.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Overdenture_2022
Record Dates: First submitted 2022-04-23; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Atrophic Maxilla; Edentulous Jaw
MeSH Terms: conditions — Atrophic Maxilla; Jaw, Edentulous

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implant assisted maxillary overdenture (Experimental): Horseshoe Maxillary Complete overdenture construction (Stabilizing and connecting the Smart Box housing)
  Interventions: Other: Implant assisted maxillary overdenture

INTERVENTIONS:
Other: Implant assisted maxillary overdenture — For each patient, an implant assisted maxillary overdenture will be fabricated using a minimally invasive flapless surgical technique with OT-Equator and Smart Box attachment

SUMMARY:
The aim of the present study is to clinically and radiographically evaluate the effect of the use of recently developed Smart Box accompanied with OT Equator attachment in retaining of the inclined implant assisted overdenture for atrophic maxilla and to compare the vertical bone changes around axial implants with OT Equator attachment and inclined implants with smart box attachment radiographically using CBCT

ELIGIBILITY:
Inclusion Criteria:

* Male patients with comparable age (30- 65 years).
* All patients should have retruded, posteriorly atrophic completely edentulous maxilla with sinus pneumatization leaving less than 7mm bone height posteriorly and a sufficient amount of bone in the inter bicuspids region.
* Opposing mandibular dentate arch including bilateral posterior teeth.
* All patients should have an adequate zone of keratinized mucosa.
* All patients should be free from any intra-oral or systemic diseases that would otherwise affect the osseointegration of dental implants.
* All patients should be well motivated, cooperative, and with adequate manual dexterity necessary to place and remove removable implant prosthesis to provide adequate oral hygiene around the endosseous implants.

Exclusion Criteria:

* Patients with flabby maxillary ridges.
* Patients who are unwilling to accept implant overdentures as a treatment modality.
* Patients with temporomandibular and neuromuscular disorders.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
change in peri-implant probing depth | Baseline, 3 months, 6 months, 9 months
  The peri-implant sulcus depth will be measured using a graduated plastic periodontal probe.
Change in Clinical Attachment level | Baseline, 3 months, 6 months, 9 months
  It is the distance from the junction implant/abutment to the most apically probable portion, in millimeters
Change in Implant Stability | at baseline and 9 months
  The Osstell unit records a numeric value of 1-100 which is referred to as the implant stability quotient (ISQ)
Change in alveolar bone level | at baseline and 9 months
  The level of alveolar bone around each abutment will be evaluated using CBCT.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt